CLINICAL TRIAL: NCT04886830
Title: Surgical Appendiceal Stump Closure - a Comparison Between Surgical Appendiceal Base Closure Methods, and Appendiceal Stump Complications.
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, yaron rudnicki, attending surgeon - surgical ward B, Meir medical center, Meir Medical Center
Other Study IDs: MeirMc - appendiceal stump
Record Dates: First submitted 2021-05-07; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: All Appendectomies Performed During the Designated Period in Single Medical Center
Keywords: laparoscopic appendectomy; appendiceal stump; endoloop

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Appendectomy performed with single endoloop to appendiceal stump: Appendectomy performed with single endoloop for closure of appendiceal stump
  Interventions: Procedure: laparoscopic appendectomy using a single endoloop for appendiceal stump closure
- Appendectomy performed with two endoloops to appendiceal stump: Appendectomy performed with two endoloops for closure of appendiceal stump
  Interventions: Procedure: laparoscopic appendectomy using two endoloops for appendiceal stump closure
- Appendectomy performed with a clip to appendiceal stump: Appendectomy performed with a clip for closure of appendiceal stump
  Interventions: Procedure: laparoscopic appendectomy using a clip for appendiceal stump closure

INTERVENTIONS:
Procedure: laparoscopic appendectomy using a single endoloop for appendiceal stump closure — laparoscopic appendectomy using a single endoloop for appendiceal stump closure before resecting the appendix
  Groups: Appendectomy performed with single endoloop to appendiceal stump
Procedure: laparoscopic appendectomy using two endoloops for appendiceal stump closure — laparoscopic appendectomy using a two endoloops for appendiceal stump closure before resecting the appendix
  Groups: Appendectomy performed with two endoloops to appendiceal stump
Procedure: laparoscopic appendectomy using a clip for appendiceal stump closure — laparoscopic appendectomy using an endoclip for appendiceal stump closure before resecting the appendix
  Groups: Appendectomy performed with a clip to appendiceal stump

SUMMARY:
comparing the rate and severity of postoperative complication after LA in regards of different appendiceal stump closure techniques. Data regarding different operative and postoperative parameters was collected from all appendectomies performed in a single medical center in Israel during the years 2010-2020.

DETAILED DESCRIPTION:
To date, laparoscopic appendectomy (LA) is still the most common surgical procedure done in an acute setting [1,2]. Most patients presenting to the ER with acute appendicitis, will undergo an appendectomy in the same hospital admission [3]. The widely practiced technique for LA, is the placement of access trocars in a proper triangulation, insufflation of the abdomen to create a pneumoperitoneum, dissecting through the mesoappendix with electrothermal devices to expose the appendiceal base, appendiceal stump closure and appendiceal resection, and finally extraction of the resected appendix [4].

There are multiple techniques to close and secure the appendiceal stump. The use of staples, clips and prepared surgical knots such as the ENDOLOOP with PDS suture is widely in use. Although requiring less manual surgical skill to use, the costs of staples and clips are higher than the prepared suture, and the use of larger trocars is obligatory [4].

Yet, data comparing the postoperative efficacy and safety of these appendiceal stump closure techniques is scarce.

The aim of this study is to compare the postoperative efficacy and safety of appendiceal stump closure techniques, and to assess their cost effectiveness.

This is a retrospective, single center study, comparing the rate and severity of postoperative complication after LA. Data regarding different operative and postoperative parameters was collected from all appendectomies performed in a single medical center in Israel during the years 2010-2020.

ELIGIBILITY:
Inclusion Criteria:

all patients over the age of 18, who underwent appendectomy between the years 2010-2020

Exclusion Criteria:

patients who did not undergo appendectomy patients who underwent appendectomy not using one of the accepted techniques do appendiceal stump closure

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients over the age of 18, who underwent appendectomy between the years 2010-2020
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
postoperative complications | 30 days
  postoperative complications such as abscess formation, perforation, need of second surgery. complications measured with clavien-dindo classification

OTHER OUTCOMES:
costs of different appendiceal stump closure techniques | 30 days
  costs of different appendiceal stump closure techniques

CONTACTS AND LOCATIONS:
Locations (1):
- Meir medical center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No